CLINICAL TRIAL: NCT03752008
Title: Preschoolers Active at Child Care
Brief Title: Preschoolers Active at Child Care (PACT)
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Pooja Tandon, Assistant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14169
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 10 childcare centers were cluster-randomized to receive either a physical activity or outdoor free play curriculum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Play (AP) (Experimental): This arm received the Active Play curriculum intervention (described in following section).
  Interventions: Behavioral: Active Play (AP)
- Outdoor Play (OP) (Experimental): This arm received the Outdoor Play curriculum intervention (described in following section).
  Interventions: Behavioral: Outdoor Play (OP)

INTERVENTIONS:
Behavioral: Active Play (AP) — This intervention focused on promoting PA in preschoolers through structured, teacher-led activities that could be incorporated into daily curriculum. Teachers attended a 3-hour workshop that included presentation and discussion of 1) the importance of daily physical activity for children's health and development, 2) teachers' beliefs and barriers to promoting PA, and 3) the Active Play! Intervention materials. Teachers were introduced to and given the Active Play! Fun Physical Activities for Young Children Book and Digital Video Disk (DVD), which promotes PA and fundamental movement skills in young children. Clips of the DVD demonstrating various activities were shown and activities were modeled. Examples of activities include jumping on bubble wrap, hula hoop limbo and an indoor obstacle course. The end of the book has a suggested curriculum that teachers could follow. Centers in the Active Play! intervention also received a set of portable toys needed for the suggested activities.
  Arms: Active Play (AP)
Behavioral: Outdoor Play (OP) — This intervention focused on promoting outdoor time in preschoolers as a means to increasing their PA, using both child initiated and teacher-led activities. The training and materials were designed to emphasize the teacher's own connection with nature, the benefits of outdoor time for children and adults, and problem solving around barriers encountered. Teachers at participating centers attended one 3-hour workshop (delivered at the childcare center) that focused on having participants recognize their own connection with the natural world and how to transmit that to the next generation. Teachers were given hats and gloves for themselves, a set of rain jackets and boots for the preschoolers, and ideas on what children could do outdoors to be active.
  Arms: Outdoor Play (OP)

SUMMARY:
The aim of this study was to develop, test, and compare two approaches to increasing physical activity (PA) and decreasing sedentary time among young children at child care centers, one which focused on a teacher-led PA curriculum (AP=Active Play!) and the other on increasing outdoor free play time (OP=Outdoor Play!).

DETAILED DESCRIPTION:
This was a matched pair cluster-randomized study in 10 child care centers. One classroom in each pair received either AP or OP, and their providers received a condition-specific 3-hour workshop. Pre- and post-intervention data were collected from classroom observation and accelerometers. Additional information about teachers' attitudes and practices was collected via pre-intervention survey.

ELIGIBILITY:
Inclusion Criteria:

* Teachers/Staff
* be a teacher/staff member in a participating childcare center
* Students
* be 3 - 5 years old
* be a full day student in the classroom where data collection was occurring

Exclusion Criteria:

-

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2014-04-24 (Actual); Study Completion 2014-04-24 (Actual)

PRIMARY OUTCOMES:
Pre to post change in preschoolers Physical Activity | baseline and 12 weeks after intervention
  Physical Activity levels measured by actigraphy monitors
Pre to post change in Physical Activity Opportunities | baseline and 12 weeks after intervention
  Minutes where students could be physically active by observation (RA observed and wrote down times for when children were engaged in various activities and categorized them as active play opportunities or non active play opportunities. Total minutes in each category were calculated.

SECONDARY OUTCOMES:
pre to post Teacher Physical Activity | baseline and 12 weeks after intervention
  Physical Activity levels measured by actigraphy monitors

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Tandon, MD MPH, Principal Investigator — Seattle Chidlren's

IPD SHARING:
Plan to Share IPD: No